CLINICAL TRIAL: NCT02948387
Title: Antibiotic Prophylaxis for Type II and III Open Fractures: a Retrospective Chart Review
Brief Title: Preventing Infections in Orthopaedic Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Olayemi Osiyemi MD (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor-Investigator, Olayemi Osiyemi MD, President, Triple O Research Institute PA
Organization: Triple O Research Institute PA (Other)
Other Study IDs: TEF-IT-40A
Record Dates: First submitted 2016-10-14; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Open Fracture
MeSH Terms: conditions — Fractures, Open

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Determine if antibiotic prophylaxis with intravenous cephalosporin and aminoglycoside in patients with Type II and II open fractures is safe and effective.

DETAILED DESCRIPTION:
1. Determine the safety and efficacy of antibiotic prophylaxis in type II and II open fractures when using IV Cephalosporin and aminoglycoside.
2. Identify the incidence of acute kidney injury.
3. Identify the type and number of associated infections
4. Identify the antibiotic resistance profile noted
5. Identify any secondary infections at sites other than the fracture site

ELIGIBILITY:
Inclusion Criteria:

* Male or Female >= 18 years old
* Patients are diagnosed with a Type II or III open fracture

Exclusion Criteria:

* Prior to treatment, report of an allergy to beta-lactam or aminoglycoside antibiotics
* pregnancy
* did not receive 72 hours of IV antibiotic prophylaxis with 1st or 2nd generation cephalosporin and either gentamicin or tobramycin
* receiving ongoing inpatient care

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are at least 18 years of age with Type II or III open fractures
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Rate of fracture site infections | 30 days
  number of infections

SECONDARY OUTCOMES:
Incidence of acute renal injury | 30 days
  number of patients with worsening renal function from baseline
type of bacteria infection | 30 days
  name of bacteria infection
resistance trend in patients with infections | 30 days
  describe the number of MDRO infections
number of secondary infections at site other than fracture sites | 30 days
  describe the number infections at secondary sites

CONTACTS AND LOCATIONS:
Overall Officials: Olayemi Osiyemi, MD, Principal Investigator — Triple O Research Institute PA
Locations (1):
- Triple O Research Institute PA, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes